CLINICAL TRIAL: NCT02427464
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of VM202 in Participants With Painful Diabetic Peripheral Neuropathy
Brief Title: Phase 3 Gene Therapy for Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMDN-003
Record Dates: First submitted 2015-04-22; First posted 2015-04-28 (Estimated); Results first posted 2022-08-22 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-08

CONDITIONS: Painful Diabetic Neuropathy; Diabetic Neuropathy, Painful
Keywords: diabetic; peripheral neuropathy; shooting pain; burning pain; pins and needles pain; foot pain; ViroMed
MeSH Terms: conditions — Diabetic Neuropathies; Peripheral Nervous System Diseases; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Engensis (VM202) (Experimental): Subjects randomized to the Engensis (VM202) treatment arm received the following intramuscular injections in each calf:
  * Day 0 - 16 injections of 0.5mL of VM202 / calf
  * Day 14 - 16 injections of 0.5mL of VM202 / calf
  * Day 90 - 16 injections of 0.5mL of VM202 / calf
  * Day 104 - 16 injections of 0.5mL of VM202 / calf
  Interventions: Biological: Engensis (VM202)
- Placebo (Placebo Comparator): Subjects in the placebo control group received the following intramuscular injections in each calf:
  * Day 0 - 16 injections of 0.5mL of VM202 vehicle / calf
  * Day 14 - 16 injections of 0.5mL of VM202 vehicle / calf
  * Day 90 - 16 injections of 0.5mL of VM202 vehicle / calf
  * Day 104 - 16 injections of 0.5mL of VM202 vehicle / calf
  Interventions: Other: placebo

INTERVENTIONS:
Biological: Engensis (VM202) — gene therapy
  Arms: Engensis (VM202)
Other: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of bilateral intramuscular injections of VM202 versus placebo in the treatment of painful diabetic peripheral neuropathy.

A total of 507 of 477 planned participants were randomized in a 2:1 ratio to one of two treatment groups. Note that 500 participants received Investigational product treatment, whereas 7 participants did not receive Investigational product treatment.

Treatments - Engensis (VM202) - 336 Engensis of 318 planned participants

Control - Placebo (VM202 vehicle) - 164 Placebo of 159 planned participants

Randomization were stratified by current use of gabapentin and/or pregabalin.

DETAILED DESCRIPTION:
Peripheral neuropathy is a serious complication of diabetes. This form of neuropathy carries a high risk of pain, trophic changes, and autonomic dysfunction. Current treatments of diabetic peripheral neuropathy are based on either pathogenetic mechanisms or symptomatic relief. A number of clinical trials have established symptomatic treatment but for pathogenetic mechanisms, the only proven treatment strategy is strict glycemic control. Clearly, it would be desirable to prevent, impede, or reverse the disrupting and often life-threatening manifestations of peripheral neuropathy by stimulating growth or regeneration of peripheral nerve axons.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years to ≤ 75 years
2. Documented history of type I or II diabetes with current treatment control (HbA1c of ≤ 10.0% at Screening) and currently on medication for diabetes (oral, injectable, and/or insulin)
3. No significant changes anticipated in diabetes medication regimen
4. No new symptoms associated with diabetes within the last 3 months prior to study entry
5. Diagnosis of painful diabetic peripheral neuropathy in both lower extremities
6. Lower extremity pain for at least 6 months
7. Visual analog scale score of ≥ 40 mm at Initial Screening (0 mm = no pain - 100 mm very severe pain)
8. Symptoms from the Brief Pain Neuropathy Screening is ≤ 5 point difference between legs at Initial Screening
9. The average daily pain intensity score of the Daily Pain and Sleep Interference Diary completed after medication wash-out is ≥ 4 with a standard deviation ≤ 2
10. The physical examination component of the Michigan Neuropathy Screening Instrument Score is ≥ 3 at Screening
11. Subjects on gabapentin (Neurontin), pregabalin (Lyrica), duloxetine (Cymbalta) for painful Diabetic Peripheral Neuropathy at study entry must be on stable regimen of these treatments for at least 3 months prior to study entry
12. If female of childbearing potential, negative urine pregnancy test at screening and using acceptable method of birth control during the study

Exclusion Criteria:

1. Peripheral neuropathy caused by condition other than diabetes
2. Other pain more severe than neuropathic pain that would prevent assessment of Diabetic Peripheral Neuropathy
3. Progressive or degenerative neurological disorder
4. Myopathy
5. Inflammatory disorder of the blood vessels (inflammatory angiopathy, such as Buerger's disease)
6. Active infection
7. Chronic inflammatory disease (e.g., Crohn's disease, rheumatoid arthritis)
8. Positive HIV or HTLV at Screening
9. Active Hepatitis B or C as determined by Hepatitis B core antibody (HBcAb), antibody to Hepatitis B surface antigen (IgG and IgM; HBsAb), Hepatitis B surface antigen (HBsAg), and Hepatitis C antibodies (Anti HCV) at Screening
10. Subjects with known immunosuppression or currently receiving immunosuppressive drugs, chemotherapy, or radiation therapy
11. Stroke or myocardial infarction within last 3 months
12. Specific laboratory values at Screening including: Hemoglobin < 8.0 g/dL, WBC < 3,000 cells per microliter, platelet count <75,000/mm3, Creatinine > 2.0 mg/dL; AST and/or ALT > 3 times the upper limit of normal or any other clinically significant lab abnormality which in the opinion of the investigator should be exclusionary
13. Ophthalmologic conditions pertinent to proliferative retinopathy or conditions that preclude standard ophthalmologic examination
14. Uncontrolled hypertension defined as sustained systolic blood pressure > 200 mmHg or diastolic BP > 110 mmHg at Screening
15. Subjects with a recent history (< 5 years) of or new screening finding of malignant neoplasm except basal cell carcinoma or squamous cell carcinoma of the skin (if excised and no evidence of recurrence for one year); subjects with family history of colon cancer in any first degree relative are excluded unless they have undergone a colonoscopy in the last 12 months with negative findings
16. Use of the following drugs / therapeutics is prohibited. Subjects may participate in the study if they are willing to discontinue use of these drugs / therapeutics 7 days prior to starting the 7 Day Daily Pain and Sleep Interference Diary. Subjects must refrain from taking these drugs or undergoing these therapies for the duration of the study

    * skeletal muscle relaxants, opioids, benzodiazepines (except for stable bedtime dose),
    * capsaicin, local anesthetic creams (except for lidocaine cream prior to intramuscular injection) and patches, isosorbide dinitrate spray,
    * transcutaneous electrical nerve stimulation (TENS), acupuncture
17. If not using gabapentin (Neurontin) or pregabalin (Lyrica), subjects must agree not to start these drugs for the first 180 days of the study. Subjects on these medications at study entry must maintain a stable dose until Day 180 of the study;
18. If not using duloxetine (Cymbalta), any antidepressants (e.g., amitriptyline and venlafaxine), any other antiepileptics (e.g., valproic acid, carbamazepine, vigabatrin), subjects must agree not to start these drugs for the first 6 months of the study.

    Subjects on these medications at study entry must maintain a stable dose until Day 180 of the study
19. Subjects requiring > 81 mg daily of acetylsalicylic acid; subjects may be enrolled if willing/able to switch to ≤ 81 mg daily of acetylsalicylic acid or to another medication
20. Subjects requiring regular COX-2 inhibitor drug(s) or non-specific COX-1/COX-2 inhibiting drugs, or high dose steroids (except inhaled steroids or ocular steroids) subjects may be enrolled if willing/able to undergo medication wash-out prior to the first dosing and to refrain from taking these drugs until Day 180 of the study
21. Major psychiatric disorder within the last 180 days that would interfere with study participation
22. Body mass index > 45 kg/m2 at Screening
23. Any lower extremity amputation due to diabetic complications
24. Use of an investigational drug or treatment in past 6 months, or prior participation in any study of Engensis (VM202)
25. Unable or unwilling to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2016-04; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Kessler, MD, Principal Investigator — Northwestern University
Locations (25):
- United States (25):
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Richard S. Cherlin, MD, Los Gatos, California
  - Northern California Research, Sacramento, California
  - Center for Clinical Research, San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Associated Neurologists of Southern Connecticut, PC, Fairfield, Connecticut
  - Innovative Research of West Florida, Clearwater, Florida
  - University of Florida McKnight Brain Institute, Gainesville, Florida
  - UF Health College of Med, Jacksonville, Jacksonville, Florida
  - Compass Research, LLC, Orlando, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center Department of Neurology, New York, New York
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Martin Foot and Ankle, York, Pennsylvania
  - Nerve and Muscle Center of Texas, Houston, Texas
  - University of Utah -Neurology, Salt Lake City, Utah
  - EVMS (Eastern Virginia Medical School), Norfolk, Virginia
  - Western Washington Medical Group, Everett, Washington
  - Rainier Clinical Research Center, Inc., Renton, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kessler JA, Shaibani A, Sang CN, Christiansen M, Kudrow D, Vinik A, Shin N; VM202 study group. Gene therapy for diabetic peripheral neuropathy: A randomized, placebo-controlled phase III study of VM202, a plasmid DNA encoding human hepatocyte growth factor. Clin Transl Sci. 2021 May;14(3):1176-1184. doi: 10.1111/cts.12977. Epub 2021 Feb 2. PMID 33465273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited using standard methods were randomized 2:1 to Engensis or Placebo and stratified by gabapentinoid use versus non-gabapentinoid concomitant medications.
Groups:
- Engensis (VM202): Participants randomized to the Engensis (VM202) treatment arm received the following intramuscular injections in each calf:
  * Day 0 - 16 injections of 0.5mL of VM202 / calf
  * Day 14 - 16 injections of 0.5mL of VM202 / calf
  * Day 90 - 16 injections of 0.5mL of VM202 / calf
  * Day 104 - 16 injections of 0.5mL of VM202 / calf
  Engensis (VM202): gene therapy
- Placebo: Participants randomized to the Placebo treatment arm received the following intramuscular injections in each calf
  * Day 0 - 16 injections of 0.5mL of VM202 vehicle / calf
  * Day 14 - 16 injections of 0.5mL of VM202 vehicle / calf
  * Day 90 - 16 injections of 0.5mL of VM202 vehicle / calf
  * Day 104 - 16 injections of 0.5mL of VM202 vehicle / calf
  placebo
Period: Overall Study
Arm/Group | Engensis (VM202) | Placebo
Started | 338 | 169
Intent-to-Treat Population | 336 | 164
Completed | 288 | 145
Not Completed | 50 | 24
Not completed — Adverse Event | 6 | 1
Not completed — Lost to Follow-up | 16 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Noncompliance | 16 | 10

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population
Groups:
- Engensis (VM202): Subjects randomized to the Engensis (VM202) treatment arm received the following intramuscular injections in each calf:
  * Day 0 - 16 injections of 0.5mL of VM202 / calf
  * Day 14 - 16 injections of 0.5mL of VM202 / calf
  * Day 90 - 16 injections of 0.5mL of VM202 / calf
  * Day 104 - 16 injections of 0.5mL of VM202 / calf
  Engensis (VM202): gene therapy
- Placebo: Subjects in the placebo control group received the following intramuscular injections in each calf:
  * Day 0 - 16 injections of 0.5mL of VM202 vehicle / calf
  * Day 14 - 16 injections of 0.5mL of VM202 vehicle / calf
  * Day 90 - 16 injections of 0.5mL of VM202 vehicle / calf
  * Day 104 - 16 injections of 0.5mL of VM202 vehicle / calf
  placebo
- Total: Total of all reporting groups
Arm/Group | Engensis (VM202) | Placebo | Total
Number analyzed (Participants) | 336 | 164 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.09) | 61.6 (9.09) | 61.0 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 45 | 188
  Male | 193 | 119 | 312
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 247 | 125 | 372
  Black or African American | 71 | 29 | 100
  Asian | 11 | 4 | 15
  American Indian or Alaska Native | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 5 | 4 | 9
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 336 | 164 | 500

OUTCOME MEASURES:

1. Primary Outcome: Change in the Average 24 Hour Pain Score From Baseline to Day 90
Description: Participants rated their 24-hour average daily pain intensity score using an 11-point numerical rating scale from 0 (no pain) to 10 (worst possible pain) in a Daily Pain and Sleep Interference Diary
Time Frame: The Pain and Sleep Interference diary was completed by participants for at least 5 assessments during a 7-day period at Screening (the mean 24-hour score was the reference/baseline score) and within 14 days prior to Day 90 visit.
Population: Overall number of Intent-to-Treat population with available data for this assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engensis (VM202) | Placebo
Number analyzed (Participants) | 312 | 154
units on a scale | -1.80 (2.05) | -1.57 (2.07)

2. Primary Outcome: Participants With at Least at 50 Percent Reduction in Average 24-hour Pain Score From Baseline to Day 90
Description: Number of participants with at least a 50 percent reduction in average 24-hour pain score, using an 11-point numerical rating scale from 0 (no pain) to 10 (worst possible pain) in the Daily Pain and Sleep Interference Diary
Time Frame: Baseline to Day 90
Population: Intent-to-Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis (VM202) | Placebo
Number analyzed (Participants) | 336 | 164
Participants | 69 | 28

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events.
Description: Number of Participants with at least one treatment-emergent adverse events.
Time Frame: Baseline to Day 270
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis (VM202) | Placebo
Number analyzed (Participants) | 332 | 161
Participants | 241 | 111

4. Secondary Outcome: Change in the Average 24-hour Pain Score From Baseline to Day 180
Description: Participants rated their 24-hour average daily pain intensity score using an 11-point numerical rating scale from 0 (no pain) to 10 (worst possible pain) in the Daily Pain and Sleep Interference Diary
Time Frame: Baseline to Day 180
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engensis (VM202) | Placebo
Number analyzed (Participants) | 336 | 164
units on a scale | -2.59 (2.38) | -2.14 (2.36)

5. Secondary Outcome: Participants With at Least a 50 Percent Reduction in Average 24-hour Pain Score From Baseline to Day 180
Description: The number of participants with at least a 50% reduction in average 24-hour pain score using an 11-point numerical rating scale from 0 (no pain) to 10 (worst possible pain) in the Daily Pain and Sleep Interference Diary
Time Frame: Baseline to Day 180
Population: Intent-to-Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis (VM202) | Placebo
Number analyzed (Participants) | 336 | 164
Participants | 113 | 42

ADVERSE EVENTS:
Time Frame: 270 days
Description: All-Cause Mortality, Serious and Other Adverse Events were monitored for the Safety Population
Arm/Group | Engensis (VM202) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/332 | 1/161
Serious Adverse Events (participants affected / at risk) | 32/332 | 16/161
Other Adverse Events (participants affected / at risk) | 237/332 | 102/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Engensis (VM202) (N=332) | Placebo (N=161)
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Infected bite (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Mononeuropathy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Influenza A virus test positive (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Engensis (VM202) (N=332) | Placebo (N=161)
Upper respiratory tract infection (Infections and infestations) | 22 | 12
Nasopharyngitis (Infections and infestations) | 17 | 4
Bronchitis (Infections and infestations) | 9 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 5
Fall (Injury, poisoning and procedural complications) | 7 | 8
Diabetic retinopathy (Eye disorders) | 7 | 10
Cataract (Eye disorders) | 9 | 3
Headache (Nervous system disorders) | 14 | 3
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Nausea (Gastrointestinal disorders) | 9 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 | 4
Oedema peripheral (General disorders) | 9 | 2
Injection Site Reaction (Grade 1 or 2) (Injury, poisoning and procedural complications) | 46 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator Agreement .....

DOCUMENTS (2):
  • Study Protocol (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT02427464/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT02427464/SAP_001.pdf